CLINICAL TRIAL: NCT06801041
Title: TRIPS - Treatment to Improve Depression and/or Anxiety Using Psilocybin-assisted Psychotherapy in Cancer Survivors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1663; NCI-2025-00634 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Depression; Anxiety; Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Psilocybin (Experimental)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will recive treatment by mouth on an outpatient basis.

SUMMARY:
This clinical research study is to learn about the feasibility, safety, and effects of psilocybin-assisted psychotherapy for cancer survivors with depression and/or anxiety.

DETAILED DESCRIPTION:
Primary Objective:

To examine the feasibility, safety, effect size estimates of psilocybin-assisted psychotherapy for cancer survivor patients with depression and/or anxiety. Feasibility will be measured as: At least 20% of eligible patients consent (inclusion rate), at least 60% of consented patients completing the two doses of treatment (treatment completion rate), and at least 80% and 65% consenting patients completing assessments at the 2- and 6-month follow-ups (adherence rates), respectively.

Secondary Objectives:

1. Determine whether psilocybin-assisted psychotherapy improves measures of quality of life (e.g., sleep, pain, functional status) and psychosocial well-being (e.g., finding meaning and post-traumatic growth), as measured by the following: PHQ-9, GAD-7, PROMIS-10, PROMIS-A, PROMIS-D, MEQ30 (mystical experience), Flourishing scale, mDES, PIQ (altered states), and Posttraumatic Growth Inventory.
2. Determine whether psilocybin-assisted psychotherapy improves functional status per clinician-rated outcome measures.
3. Measure the change in inflammatory markers (IL6, TNF, and CRP) and in frequency and activation status of peripheral immune cell populations assessed by immune monitoring through flow cytometry.
4. Examine changes in central nervous system plasticity through the use of fMRI, specifically changes in 5-HT2A-rich and higher-order functional networks, as well as a global increase in brain network integration.
5. Evaluate the Impact on MDASI measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have solid or hematological malignancy that does not involve the brain.
2. Documentation of current malignancy that was treated and the patient has no evidence of disease in the previous 6 months
3. Age ≥ 18 years.
4. Have a DSM-V psychiatric diagnosis, as determined by the SCID (Structured Clinical Interview for DSM), of one or more of the following Axis I psychiatric disorders that is judged to have been precipitated by the psychological stress of the cancer diagnosis: Generalized Anxiety Disorder; Acute Stress Disorder; Posttraumatic Stress Disorder; Major Depressive Disorder, Dysthymic Disorder; Adjustment Disorder with Anxiety; Adjustment Disorder with Depressed Mood; Adjustment Disorder with Mixed Anxiety and Depressed Mood; Adjustment Disorder with Disturbance of Conduct; Adjustment Disorder with Disturbance of Emotions and Conduct. Psychiatric diagnoses are determined by. an MD Anderson licensed healthcare provider with graduate-level profession training and clinical experience in psychotherapy, licensed to practice independently.
5. Have an ECOG performance status of 0, 1, or 2.
6. Must have no major cognitive impairment and be oriented to person, place, and time (e.g. mini mental exam).
7. Must demonstrate willingness to travel to MD Anderson Cancer center for all treatment and follow-up sessions, as well as consent to complete all evaluation instruments and assessments.
8. Agree to abstain from any nicotine products for at least 8 hours prior to fMRI performance.
9. Refrain from any psychoactive drugs (including alcohol) for 48 hours prior to psilocybin sessions and must refrain from psychoactive drugs 12 hours after psilocybin sessions. Must consent to urine drug screen (UDS) which will be given before receiving psilocybin. Participants with positive drug test will be retested (UDS) after 6 weeks and included if the repeated UDS is negative. Patient tested positive for a prescribed substance are eligible. Patient failing on the 2nd test (UDS) will be excluded.
10. Must be free from any regularly scheduled psychotropic (antidepressant/anxiolytic class) medications for a minimum of 2 weeks prior to study. Intermittent or PRN use of short-acting anxiolytics or and anti-nausea medications (e.g., ondansetron) may be permitted as defined below in exclusionary criteria). Ondansetron could be taken but must be stopped at least 24 hours before psilocybin administration.
11. Inhibitors of monoamine oxidase, UGT1A9, 1A10, and aldehyde or alcohol dehydrogenase should be discontinued 5 half-lives prior to active dose of psilocybin.
12. Eligible subjects will have a third-party transportation by a licenses driver (e.g. friend, family or a driver) after the psilocybin session is complete. If a driver is used, a friend or family member must accompany them in the vehicle home
13. Fluent in Englishria). Ondansetron could be taken but must be stopped at least 24 hours before psilocybin administration.

Exclusion Criteria:

1. Clinically significant suicidality or high risk of completed suicide defined as:

   i. Answer 'Yes' to C-SSRS Suicidal Ideation items 4 or 5 within the last 2 months at Screening or 'since last visit' at Baseline ii. Report having had any C-SSRS Suicidal Behavior item within the past 12 months at Screening or 'since last visit' at Baseline, as defined by 'Yes' to any of the following on the C-SSRS: actual attempt, interrupted attempt, aborted attempt, or preparatory acts iii. Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self injurious behavior
2. History of bipolar disorder, psychosis (including a history of schizophrenia).
3. Functionally limiting comorbid conditions such as second primary malignancies in CNS or chest, and history of total laryngectomy or total glossectomy precluding them from communicating.
4. The effects of psilocybin on the developing human fetus are unknown. For this reason, pregnant women will be excluded (Urine test for screening), women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstaining from intercourse with the opposite sex) prior to study entry and for the duration of study participation. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
5. Persons with first-degree relatives who have schizophrenia or other psychotic disorders, or bipolar I or II disorder diagnosed by a qualified mental health professional.
6. Documentation of current malignancy that is being treated with palliative intent.
7. Vulnerable populations, including children and cognitively impaired patients, will not be enrolled in this study.
8. Patients with brain metastases.
9. Risk for hypertensive crisis defined as Screening, Baseline, and Medication Session (day of dosing, prior to dosing) Blood Pressure >blood pressure >180/120mmHG, HR >110 bpm . Of note, we will repeat vital signs for subjects with high initial reading and average three readings to determine eligibility criteria in such cases to account for normal variability in vital sign and "white coat hypertension."
10. Unstable medical conditions or serious abnormalities of complete blood count, chemistries, or ECG that in the opinion of the study physician would preclude safe participation in the trial. Some examples include:

    i. Uncompensated congestive heart failure ii. Clinically significant arrhythmias (e.g., ventricular fibrillation, torsades) or clinically significant ECG abnormality (i.e., QTC interval > 450) iii. Recent acute myocardial infarction or evidence of ischemia iv. Malignant hypertension v. Congenital long QT syndrome vi. Acute renal failure vii. Severe hepatic impairment viii. Respiratory failure
11. Significant central nervous system (CNS) pathology. Some examples include:

    i. Primary or secondary cerebral neoplasm on imaging ii. Epilepsy and any history of seizure (regardless of if related to epilepsy) except for a one-time febrile seizure in childhood iii. History of stroke in the past 3 years iv. Untreated cerebral aneurysm v. Dementia vi. Ongoing delirium in which subjects would not have the capacity to participate in the study.

12 a. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation. Examples include: i. Agitation ii. Violent behavior b. Active substance use disorders (SUDs) defined as: DSM-5 criteria for moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine) within the past year c. Extensive use of serotonergic hallucinogens (e.g., LSD, psilocybin) defined as: i. Any use in the last 12 months ii. >22 lifetime uses d. History of hallucinogen persisting perception disorder (HPPD) e. Concurrent Medications i. Antidepressants ii. Centrally-acting serotonergic agents (e.g., MAO inhibitors) iii. Antipsychotics (e.g., first and second generation) iv. Mood stabilizers (e.g., lithium, valproic acid) v. Aldehyde dehydrogenase inhibitors (e.g., disulfiram) vi. Significant inhibitors of UGT 1A0 or UGT 1A10 vii. serotonin-acting dietary supplements (such as 5-hydroxytryptophan or St. John's wort) viii. efavirenz f. Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP), and Tetrahydrocannabinol (THC).

i. Note: Prescribed opiate medications (e.g., cancer-related pain) will be allowed to continue through the study period for participants who have been on a stable dose of such medicine for at least 1 month prior to Screening, as determined during review of concomitant medications.

ii. Note: Prescribed benzodiazepine medications and nonbenzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications.

iii. Note: Participants using cannabis, including legal cannabis, for any purposes must agree to refrain from use beginning at Screening, as confirmed with a negative Baseline drug test, and through to the end of the study.

iv. Note: Participants using prescribed psychostimulants (amphetamines and Ritalin), must agree to refrain from use 72 hours prior to dosing and until 12 hours after dosing.

g. Have a psychiatric condition judged to be incompatible with establishment of rapport with the study therapists or safe exposure to psilocybin.

h. Have any psychological or physical symptom, medication or other relevant finding prior to randomization, based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.

i. Have an allergy or intolerance to any of the materials contained in the drug product.

j. Be enrolled in another clinical trial assessing intervention(s) for anxiety, depression, and/or existential distress (e.g., pharmacologic or psychotherapeutic interventions).

13. Patients with non-fMRI compatible implants will be eligible but will not have fMRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Moran Amit, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M. D, Anderson Cancer Center Website — http://www.mdanderson.org